CLINICAL TRIAL: NCT02480543
Title: Different Routes of Misoprostol for Same-day Cervical Preparation Prior to First Trimester Surgical Abortion: a Randomized Controlled Trial
Brief Title: Different Routes of Misoprostol Prior to First Trimester Surgical Abortion
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Hadas Ganer Herman, MD, Wolfson Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0085-15-WOMC
Record Dates: First submitted 2015-06-20; First posted 2015-06-24 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Abortion, Induced
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- PO Misoprostol (Active Comparator): Cervical preparation with per-os (PO) Misoprostol 400 mcg 2-4 hours prior to curettage
  Interventions: Drug: Misoprostol (cytotec)
- PV Misoprostol (Active Comparator): Cervical preparation with per-vagina (PV) Misoprostol 400 mcg 2-4 hours prior to curettage
  Interventions: Drug: Misoprostol (cytotec)
- Buccal Misoprostol (Active Comparator): Cervical preparation with buccal Misoprostol 400 mcg 2-4 hours prior to curettage
  Interventions: Drug: Misoprostol (cytotec)

INTERVENTIONS:
Drug: Misoprostol (cytotec)

SUMMARY:
A randomized clinical trial to assess the effectiveness of same-day cervical preparation with oral, buccal or vaginal Misoprostol, given 2-4 hours prior first trimester curettage.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted for elective first trimester abortion (termination of pregnancy/ missed abortion) at Wolfson Medical Center, gestational age <13+0 weeks
* Written consent supplied

Exclusion Criteria:

* Contraindications to prostaglandin treatment (severe asthma, glaucoma, severe cardiac disease, renal failure)
* Prostaglandin allergy
* Genital infection
* Space-occupying lesion in the endocervical canal
* Prior cervical surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Preoperative cervical width in centimeters | intraoperative
  • Initial cervical dilatation assessed by performing cervical dilatation , beginning with a number 10 Hegar dilator and subsequently inserting smaller Hegar dilators until the dilator can pass through the internal os without resistance. The largest one to pass will consist the initial cervical width.

SECONDARY OUTCOMES:
Time required to achieve cervical dilatation | intraoperative
  The time in minutes required for dilatation up to a number 10 Hegar
Ease of cervical dilatation | intraoperative
  The subjective ease of cervical dilatation recorded by the surgeon on a 5-point Likert scale (1-very difficult, 5- very easy
Patient preference | baseline
  Patient acceptability of the administration of medication on a 5-point Likert scale (1-very uncomfortable, 5-very comfortable)
Adverse effects of medication | baseline
  Self reported misoprostol-associated adverse effects before the procedure (such as nausea, vomiting)
Surgical complications | intraoperative
  Complications arising during surgery (perforation, cervical laceration, excess bleeding)

CONTACTS AND LOCATIONS:
Overall Officials: Hadas Ganer Herman, MD, Principal Investigator — Edith Wolfson Medical Center
Locations (1):
- Edith Wolfson Medical Center, Holon, Israel

REFERENCES:
- [Derived] Ghosh J, Papadopoulou A, Devall AJ, Jeffery HC, Beeson LE, Do V, Price MJ, Tobias A, Tuncalp O, Lavelanet A, Gulmezoglu AM, Coomarasamy A, Gallos ID. Methods for managing miscarriage: a network meta-analysis. Cochrane Database Syst Rev. 2021 Jun 1;6(6):CD012602. doi: 10.1002/14651858.CD012602.pub2. PMID 34061352